CLINICAL TRIAL: NCT01482078
Title: Prospective Observational Study, Maternal Effects of Magnesium Sulphate for Neonatal Neuroprotection in Women Having Cesarean Section Under Neuraxial Anesthesia
Brief Title: Magnesium for Neonatal Neuroprotection and Mothers
Acronym: MnMs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, James Brown, Principle Investigator, University of British Columbia
Other Study IDs: H11-02970
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Premature Birth; Sedation During Labor and Delivery; Complications, Pulmonary; Respiratory Depression
Keywords: Magnesium Sulphate; Neuroprotection; Neuraxial Anesthesia; Sedation; Respiratory function; Cesarean Section; Obstetrical Anesthesia
MeSH Terms: conditions — Premature Birth; Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Receive MgSO4 infusion: Parturients who present to the hospital at less than 34 weeks gestational age with potential pre-term labor, pre-term rupture of membranes or intrauterine growth restriction
- Do not receive MgSO4 infusion: We will approach a control group of subjects: i.e. parturients undergoing cesarean section (elective or emergency) with neuraxial anesthesia.
  We will seek to ensure that the control group is similar to the study group with respect to the following parameters:
  * Number of singleton or multiple pregnancy
  * Parity of parturients
  * Anesthetic technique (spinal or epidural)
  * Time of cesarean section (08:00-19:59 or 20:00 to 07:59) Once informed consent is obtained these subjects will be treated identically to the study group in terms of anesthetic management and data collection.

SUMMARY:
Magnesium is a treatment for mothers to protect brains of babies born early. This study investigates combined effects of magnesium and spinal or epidural anesthesia on mothers having cesareans.

The investigators will use a scoring system to measure sedation and devices that subjects breath in and out of to measure breathing strength.

The investigators hypothesize the combination of magnesium and anesthesia will reduce breathing strength and cause sedation.

This is an observational study comparing those having magnesium and anesthesia with those just having anesthesia. Routine medical care will not be altered.

Results will hopefully allow anesthesiologists to provide better patient care.

DETAILED DESCRIPTION:
1. Purpose

   Neonatal neuroprotection is a new indication for magnesium. Meta-analysis of the available literature suggests beneficial neonatal outcomes, but the direct effects on maternal health have not been studied. Unwanted effects of magnesium therapy such as sedation and respiratory insufficiency may be potentiated by neuraxial anesthesia placing the mother at risk of morbidity.
2. Hypothesis or Aim

   Magnesium causes sedation and muscle weakness, which potentiates effects of neuraxial anesthesia, increases respiratory insufficiency, reduces cough effectiveness and increases pulmonary aspiration risk. We hypothesise that compared to the control group, the group receiving magnesium will have a reduced Maximal Expiratory Pressure (MEP) by ≥15 cmH2O, or a 10% higher incidence of a composite sedation score ≤ 3.
3. Justification for the study

   There is strong evidence in the medical literature to support the current guidelines and practice to treat parturients presenting for pre-term delivery, less than 34 weeks with magnesium. The presumed benefits are a reduction in the incidence and functional motor deficit from cerebral palsy, and possibly reduction in infant mortality. Treatment with magnesium represents the current accepted practice and level of care.

   Approximately 50% of these pre-term patients will require neuraxial anesthesia to enable cesarean section, using either intrathecal or epidural techniques. There are potential cumulative side effects from neuraxial anesthesia and magnesium but no studies have been done to examine this.

   Safety of magnesium in parturients has been demonstrated. The effects of magnesium are known as it is an established therapy in the management of pre-eclampsia. The consequences of neuraxial anesthesia are also well documented. This is a prospective observational study investigating the combined effects of magnesium administration and neuraxial anesthesia. Of particular interest are effects that may place the parturient at increased risk of complications, which need active assessment and management by anesthesiologists e.g. risks of pulmonary aspiration as a result of sedation, vomiting or reduced cough effectiveness.

   In addition to the effects of magnesium and neuraxial anesthesia, ventilatory mechanics in the parturient are further compromised by:
   * the effects of the gravid uterus, displacing the diaphragm and altering the subcostal angle.
   * supine positioning on the operating table impeding ventilation because of the gravitational effect on abdominal contents.
   * the practice of "skin-to-skin" in the operating room, sitting baby on the patient's chest and mechanically impeding respiratory effort.

   Although we are interested in potential complications due to the use of magnesium in conjunction with neuraxial anesthesia, there are potential advantages of magnesium for the mother, especially with epidurals, including a reduction in shivering and improved quality of analgesia.
4. Research Method

This is a prospective, observational study with a comparison control group.

Our target population is women delivering by cesarean with neuraxial anesthesia at BC Women's Hospital. The study group includes those women <34 weeks who are receiving magnesium for neonatal neuroprotection, and the control group includes those >34 weeks who are not receiving magnesium for neonatal neuroprotection.

We propose to study a convenience sample over a 5-month period. In the last 3 years at BC Women's Hospital there have been a mean of 243 deliveries per year at less than 34 weeks and 128 of these are by cesarean section. Over a 5-month period with an average number of presentations it would be theoretically possible to recruit 50 patients.

We realistically expect to recruit 20 patients to the study group. A larger pool of patients is available for the control group and we will aim to recruit the number as directed by the power calculation.

Sample Size and statistical analysis:

The sample size has been chosen for the primary outcome of MEP, to determine a minimum difference in means of 15 cmH20, with an alpha or 0.05 and power of 0.8. The two-sample t-test will be used to analyse normally distributed data (e.g. MEP, MIP, FVC). Chi-squared tests will be used to compare categorical variables between the groups (e.g. composite sedation score OAA/S ≤3 or >3). If there is a significant between group difference we plan to undertake regression analysis to identify independently contributing effects after taking into account demographic factors.

It is hoped that the study will be beneficial in increasing understanding of potential effects of combining magnesium and neuraxial anesthesia in the obstetric population presenting for pre-term cesarean section. Highlighting any potential risks and improving patient safety in the future. This study will to a certain extent also be hypothesis generating in nature.

ELIGIBILITY:
Inclusion Criteria:

* Delivering by cesarean section at less than 34 weeks gestational age (maximum 33 weeks and 6 days).
* ≥19 yr
* Singleton or multiple pregnancy

  o There is potentially greater intra-abdominal pressure associated with multiple pregnancies, which may affect anesthetic block height by increasing blood volume in epidural blood vessels. It may also increase the risk of basal atelectasis and will affect respiratory mechanics to a greater extent. We plan to undertake sub-group analysis to test this effect.
* Primiparous or multiparous
* English-speaking
* Undergoing cesarean section with neuraxial anesthesia (intrathecal, epidural or combined spinal epidural [CSE]).

  * Parturients response may not be identical to the different neuraxial techniques, e.g. the degree of respiratory motor blockade exhibited or onset of opioid effect. Therefore we plan to undertake sub-group analysis to test this effect.

Exclusion Criteria:

* Illegal, non-prescription drug use within the last year
* Psychiatric disorder treated with medication within the last year

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstetric patients planning to deliver at British Columbia's Women's Hospital
  * MgSO4 infusion cohort
    -Eligible parturients at less than 34 weeks gestational age with potential pre-term labor, pre-term rupture of membranes or intrauterine growth restriction.
  * Non-MgSO4 infusion cohort -We will approach a control group of subjects: i.e. parturients undergoing cesarean section (elective or emergency) with neuraxial anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01-26 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Maximal Expiratory Pressure | 3 minutes for each of 5 tests over 2 hours
  We consider 15 cmH20 difference in MEP to be clinically significant.
Composite sedation score | 30 seconds for each of 6 tests over 2 hours
  A composite score of ≤3 (at any data collection point). This implies one of the following criteria:
  * Subject responds only after name is spoken loudly or repeatedly
  * Speech is slurred or slow
  * Marked relaxation of facial expression
  * Both eyes are glazed with marked ptosis.
  We judge this degree and incidence of sedation to be clinically significant. It would certainly be sufficient to interfere with maternal interaction with the newborn, would likely affect maternal memory of the event, and would place the mother at risk of potential airway compromise and respiratory insufficiency.

SECONDARY OUTCOMES:
To compare the following respiratory measurements | 3 minutes for each of 5 tests over 2 hours
  * oxygen saturation ≤95% (% of patients)
  * ETCO2 increase of ≥5mmHg from baseline (% of patients)
  * MEP ≤ 60cmH20 (% of patients)
  * MIP 30% decrease from baseline (% of patients)
  * Forced Vital Capacity (FVC) decrease ≥30% from baseline (% of patients)
To compare the following sedation measurements | 30 seconds for each of 6 tests over 2 hours
  * lowest sedation score <4 (% of patients)
  * sedation score decrease of >1 from baseline (% of patients) • nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: James Brown, MB BCh, Principal Investigator — BC Women's Hospital, University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada